CLINICAL TRIAL: NCT04011124
Title: A Single Center, Single Arm, Open and Fixed Sequence Study to Investigate the Pharmacokinetic Effects of Rifampicin on Fluzoparib in Healthy Male Subjects
Brief Title: A Drug-drug Interaction Trial of Rifampicin Pharmacokinetics Effect on Fluzoparib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FZPL-I-110
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — fluzoparib; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rifampicin + Fluzoparib (Experimental)
  Interventions: Drug: Fluzoparib; Drug: Rifampicin

INTERVENTIONS:
Drug: Fluzoparib — single dose on Day 1 and Day 12
Drug: Rifampicin — QD on Day 5-14 for 10 days

SUMMARY:
The primary objective of the study was to assess the effect of repeated oral doses of Rifampicin on the pharmacokinetic profile of a single dose of Fluzoparib.

The secondary objective of the study was to assess the safety of Fluzoparib given alone versus Fluzoparib coadministered with Rifampicin.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial and fully understand the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Age on the date of signing the informed consent form is 18 to 50 years old (including both ends) and is limited to male subjects only;
4. Male subjects are willing to have no birth plans in the next 6 months and voluntarily take effective contraception;
5. The fasting weight is not less than 50kg, and the body mass index (BMI) is in the range of 18 kg/m2 to 28 kg/m2 (including both ends);
6. Health status: no medical history of heart, liver, kidney, digestive tract, nervous system, mental abnormalities and metabolic abnormalities;
7. Accepted physical examination results (vital signs, physical examination) and routine laboratory examination (blood routine, blood biochemistry, urine routine, etc.), 12-lead ECG, X-chest, abdominal B-ultrasound, etc. or no clinical significance if abnormal.
8. Creatinine clearance (CLCr) ≥ 80 mL/min, and creatinine is less than or equal to the upper limit of normal

Exclusion Criteria:

1. Participate in blood donation within 3 months before screening and donate blood volume ≥400mL or blood loss ≥400mL, participate in blood donation within 1 month before screening and donate blood volume ≥200mL or blood loss ≥200mL, or receive blood transfusion;
2. Allergic constitution, including a history of severe drug allergy or drug allergy; a history of allergies to fluzoparib capsule or its excipients;
3. with drug and/or alcohol abuse history, or alcohol, nicotine and drug screening positives, or drug abuse in the past five years or used drugs 3 months before the trial; and could not prohibit smoking and alcohol during the trial period ;
4. with medical history of cardiovascular disease such as myocarditis, coronary heart disease, pathological arrhythmia, and stroke;
5. Pulmonary diseases, including invasive lung disease, pneumonia, dyspnea, etc.;
6. Chronic kidney disease, renal insufficiency, history of renal anemia;
7. have a history of dysphagia or any history of gastrointestinal disease that affects drug absorption;
8. any uncontrolled peptic ulcer, colitis, pancreatitis, etc.;
9. Anyone who has undergone any surgery within the first 6 months of screening; has undergone any surgery that affects gastrointestinal absorption (including gastrectomy, bowel resection, stomach reduction, etc.);
10. with acute disease that has been clinically determined by the investigator occurred within 1 month before screening;
11. Other important organ diseases such as the nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolic and musculoskeletal system with clear medical history (such as uncontrolled diabetes, high blood pressure, etc.), enabling investigators considered unsuitable for participation in the study;
12. Those who have taken any clinical trial drugs within 3 months;
13. Take any drug that affects liver metabolism within 28 days before taking the investigational drug;
14. Take any prescription or over-the-counter medication within 14 days before taking the investigational drug;
15. Take any vitamin products or herbs within 14 days before taking the investigational drug;
16. Clinical laboratory tests are abnormal and clinically significant, or other clinical findings indicate the following diseases, including but not limited to gastrointestinal, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular disease;
17. combined with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive) or combined with syphilis infection;
18. The subject refused to discontinue any beverage containing methylxanthine, such as caffeine (coffee, tea, cola, chocolate, etc.) or alcoholic beverages or any juice, 48 hours before the investigational drug was administered until the end of the study;
19. Strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, excretion, etc.;
20. The investigator believes that the subjects are not eligible to participate in this trial.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Fluzoparib | Day 1 to Day 15
Area under the plasma concentration versus time curve (AUC) of Fluzoparib | Day 1 to Day 15

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 22
  Laboratory indicators, 12-lead electrocardiogram (ECG), physical examination, vital signs, adverse events (NCI-CTC AE 5.0), etc.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China